CLINICAL TRIAL: NCT03329313
Title: Effects of Variation of Sodium Dialysate in ICU Acute Kiney Injury
Brief Title: Effects of Variation of Sodium Dialysate in ICU
Acronym: NADIRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL16_0254; 2017-A01704-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-09-07; First posted 2017-11-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Renal Replacement Therapy
Keywords: Intensive care unit; SLEDD-f; intermittent hemodialysis/diafiltration
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Masking Description: simple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low sodium concentration (Active Comparator): Concentration of sodium in dialysate at 140 mmol/l ( Lowering sodium concentration dialysate)
  Interventions: Drug: Lowering sodium concentration dialysate
- High Sodium Concentration (Sham Comparator): Concentration of sodium in dialysate at 145 mmol/l (Highing sodium concentration dialysate)
  Interventions: Drug: Highing sodium concentration dialysate

INTERVENTIONS:
Drug: Lowering sodium concentration dialysate — Concentration of sodium in dialysate at 140 mmol/l
  Other Names: Concentration of sodium in dialysate at 140 mmol/l
  Arms: Low sodium concentration
Drug: Highing sodium concentration dialysate — Concentration of sodium in dialysate at 145 mmol/l
  Other Names: Concentration of sodium in dialysate at 145 mmol/l
  Arms: High Sodium Concentration

SUMMARY:
Intermittent hemodialysis/diafiltration is a current renal replacement therapy (RRT) institued for ICU patients with AKI. For a better clinical tolerance, iinternational guidelines advise to use cold dialysate, increase duration session, decrease blood and dialysate flows, and increase level of sodium dialysate concentration (≥ 145mmol/l). Indeed, the use of a Na concentration dialysate > 145 mmol/l improves intradialytic hemodynamic tolerance but it may also induce fluid overload by the transfert of sodium from the dialysate compartment to the blood. Yet, fluid overload has been strongly associated with mortality in critically ills. The investigators hypothesized that the use of a level in sodium dialysate at 140 mmol/l with slow low efficiency daily dialysis-filtration (SLEDD-f) will permit a fair intradialytic hemodynamic tolerance without the adverse effect of intradiaclytic Na loading from the dialysate. Two randomized groups of ICU AKI patients treated by SLEDD-f will be compared in terms of intradialytic hemodynamic tolerance and overload accordong to 140 or 145 mmol/l of Na in the dialysate

DETAILED DESCRIPTION:
Acute kidney injury (AKI) requiring renal replacement therapy (RRT) occurs in 5 to 6% of critically ill patients and is associated with high mortality and significant health resource utilization. Modalities of RRT currently available include intermittent hemodialysis/diafiltration (IHD/F) and continuous renal replacement therapies. Continuous veno-venous therapies have gained wide application in ICUs, often supplanting IHD because of the belief that it is better tolerated in hemodynamically unstable patients. Previous reports have shown however that intermittent therapies may permit similar hemodynamic tolerance but with specific parameters including dialysate composition. Consequently, international guidelines suggest in ICU AKI the use of intermittent modalities with the use of cold dialysate, increased duration session, decreased blood and dialysate flows, and high level of sodium dialysate concentration (≥ 145mmol/l). Increasing the level of sodium dialysate concentration improves obviously the hemodynamic tolerance but may also result in inflated extracellular volume and fluid overload secondary to sodium transfert from the dialysate compartment to the blood. There is a body of evidence that fluid overload may be harmful to the critically ill, has an adverse impact and worsens outcome.

The aim of the study is therefore to compare perdialytic hemodynamic tolerance and fluid overload after 7 days of SLEDD-f using 2 sodium dialysate concentrations -140 vs 145 mmol/l- in ICU AKI patients. The investigators also planned to evaluate and compare mean ultrafiltration rate by patient, total duration of RRT, fluid overload at RRT weaning, ICU length of stay and 28 days ICU mortality using these 2 levels of sodium dialysate concentration.

Methods: This randomised, single center, prospective and non blinded study is being held in medical ICU at Lapeyronie University Hospital of Montpellier.

Patient more than 18 years old, admitted to the ICU for AKI requiring RRT and with a sSofa score > 5 will be included.

RRT will be an on line predilution SLEDD- with the following parameters: blood flow 200ml/min, dialysate flow 200ml/min, infusate flow 60ml/min, temperature 36°C, membrane polysulfone Fx80. An hemodynamic monitoring will be performed at each dialysis session. Weight, daily input and output and extracellular volume will be monitored during ICU stay.

According to the sodium concentration dialysate: 140 or 145 mmol/l, 2 groups will be randomized and compared regarding to hemodynamic tolerance, fluid overload and outcome.

Hypothesis: The use of a sodium dialysate concentration at 140 mmol/l with SLEDD-f will induce a similar intradialytic hemodynamic tolerance as compared to a Na dialysate at 145 mmmol/l but with a decrease at around 4% of fluid overload.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years old
* Acute kidney injury requiring renal replacement therapy
* Dialysis type: on line sustained low efficiency dialy dialysis -filtration
* SOFA score > 5
* Sodium serum level between 135 and 145mmol/l

Exclusion criteria:

* Chronic kidney disease stade IV ou V
* Obstrutive acute kidney injury
* Renal tansplantation in the year before ICU admission
* Moribund with risk of death in the 48 hours
* Vulnerable persons or protected persons
* Pregnant or breastfeeding mother

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Fluid overload | 7 days after the initiation of renal replacement therapy
  Daily weight measure from the initiation to the weaning of RRT. Daily monitoring of inpout and output.
Fluid overload | day 28
  Daily weight measure from the initiation to the weaning of RRT.

SECONDARY OUTCOMES:
Intradialytic hemodynamic tolerance | during the requiring renal replacement therapy (RRT)
  Intradialytic hemodynamic tolerance
Mean ultrafiltration rate by patient/ session | 1 day
  Appreciation of ultrafiltration rate for each patient and for each RRT session for all the renal replacement therapy. Calcultate the mean ultrafiltration rate by patient. Daily Weight measurement before and after each RRT session and daily
Fluid overload | 1 day
  Fluid overload after RRT weaning and ICU stay.
Total duration of RRT | 1 day
  Total duration of RRT at end of hospitalization
length of stay | 1 day
  Length of stay in the service at hospital discharge
Mortality rate | 28 days of admission
  Mortality rate at 28 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: vincent BRUNOT, MD, Principal Investigator — University Hospital, Montpellier; aurèle BUZANCAIS, MD, Study Director — UHNIMES
Locations (1):
- Uhmontpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC